CLINICAL TRIAL: NCT00408317
Title: A Multicenter, Randomized, Double-Blind, Crossover Study to Compare the Safety and Efficacy of Ultrase® MT20 to Placebo for the Correction of Steatorrhea in Patients With Cystic Fibrosis (CF)
Brief Title: Safety and Efficacy Study of ULTRASE® MT20 in Participants With Cystic Fibrosis (CF) and Exocrine Pancreatic Insufficiency (PI)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: UMT20CF05-01
Record Dates: First submitted 2006-12-04; First posted 2006-12-06 (Estimated); Results first posted 2014-03-12 (Estimated); Last update posted 2017-03-16 (Actual); Status verified 2017-02

CONDITIONS: Cystic Fibrosis; Exocrine Pancreatic Insufficiency
Keywords: Cystic Fibrosis; Exocrine Pancreatic Insufficiency; Ultrase® MT20
MeSH Terms: conditions — Cystic Fibrosis; Exocrine Pancreatic Insufficiency

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ultrase® MT20 (Experimental)
  Interventions: Drug: Ultrase® MT20
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ultrase® MT20 — Ultrase® MT 20 capsules containing enteric-coated minitablets orally daily at a dose stabilized during the first stabilization period (4 days), as per investigator's discretion, for 6 to 7 days in either first intervention period or second intervention period.
  Other Names: Pancreatic enzyme product
  Arms: Ultrase® MT20
Drug: Placebo — Placebo matched to Ultrase® MT 20 capsules orally daily for 6 to 7 days in either first intervention period or second intervention period.
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the safety and efficacy of Ultrase® MT20 compared to placebo for the correction of fat and protein malabsorption in participants with cystic fibrosis (CF) and exocrine pancreatic insufficiency (EPI). This study is sponsored by Aptalis Pharma (formerly Axcan).

DETAILED DESCRIPTION:
This is a Phase III, multicenter, randomized, double-blind, two-period cross-over, placebo-controlled study designed to compare the efficacy and safety of Ultrase® MT20 to placebo in participants with CF and pancreatic insufficiency. The study consists of a screening period (up to 11 days) and two treatment periods (6-7 days). During screening period participants will be treated with open-label Ultrase® MT18 or MT20. Each treatment period will be preceded by a stabilization period (4 days) and the two treatment periods are separated by a break period (3-6 days). A safety follow-up visit will be performed 7-10 days after discharge from the last treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Participants or their legally authorized representative must understand the nature of the study and sign an informed consent or assent form along with a parental form
* Participants must have a confirmed diagnosis of CF based on 1 or more clinical features consistent with the CF phenotype, and one of the following:

  * A genotype with 2 identifiable mutations consistent with CF
  * A sweat chloride test greater than 60 millimole per liter (mmol/L) by quantitative pilocarpine iontophoresis
* Participants must have PI as demonstrated by a fecal elastase-1 (FE-1) concentration less than 100 microgram per gram (mcg/g) of stools (ScheBo test) and must require pancreatic enzyme supplementation
* Participants must be clinically stable as evidenced by medical and medication history, baseline physical examination including vital signs and laboratory analyses
* Participants must be 7 years and older
* Participants must have an adequate nutritional status based on the following body mass index (BMI):

  * Participants 7 to 20 years old must have a BMI greater than or equal to fifth percentile
  * Female participants greater than 20 years old must have a BMI greater than or equal to 16
  * Male participants greater 20 years old must have a BMI greater than or equal to 16.5
* Participants must be on an optimal clinical dose of pancreatic enzymes (Ultrase® MT18 or MT20 or other pancreatic enzymes preparations including Ultrase® MT12) prior to entry in the study, and must tolerate this medication in the opinion of the investigator
* Participants must be able to swallow capsules and must be able to eat a high fat diet calculated as 2 gram (± 15%) fat per kilogram body weight per day
* Participants must be, in the opinion of the investigator, able and willing to complete this study
* Female participants must be premenarcheal, surgically sterile or postmenopausal for at least 12 consecutive months. Otherwise, the women of childbearing potential (WOCBP) must not be pregnant and must have practiced an acceptable method of contraception for at least one month prior to the study entry

Exclusion Criteria:

* Participants with a known contraindication, sensitivity or hypersensitivity to Ultrase or any porcine protein
* Participants with a known allergy to the food drug and cosmetic (FD&C) Blue No. 2 dye indicator (stool marker)
* Participants not willing to stop the prohibited medications or products at study entry and throughout the study
* Participants who are using narcotics
* Participants who are using bowel stimulants and/or laxatives on a regular basis
* Participants with acute pancreatitis or acute exacerbation of chronic pancreatic disease
* Participants with an acute pulmonary infection
* Participants with a history of bowel resection
* Participants suffering from any dysmotility disorders
* Participants with chronic or severe abdominal pain
* Participants receiving enteral tube feeding and not willing to stop during the course of the study
* Participants known to have a significant medical disease that would compromise their welfare or confound the study results
* Participants with a history of or a current diagnosis of clinically significant portal hypertension
* Participants who have a condition known to increase fecal fat loss including celiac's disease, biliary cancer, biliary stricture, cholelithiasis, Crohn's disease, pancreas cancer, radiation enteritis, tropical sprue, Whipple's disease, lactose intolerance, pseudomembranous colitis
* Participants with a current diagnosis or a history of complete distal intestinal obstruction syndrome (DIOS) in the past 6 months; or, participants who had 2 or more episodes of DIOS in the past year
* Participants with poorly controlled diabetes to the investigator's opinion
* Female participants who are pregnant or lactating
* Participants who received an investigational drug within 30 days prior to entry into the study

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2006-11; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aptalis Medical Information, Study Director — Forest Laboratories
Locations (4):
- United States (4):
  - DeVos Children's Hospital, Grand Rapids, Michigan
  - Rainbow Babies & Children's Hospital, Cleveland, Ohio
  - Pennsylvania State University, The Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - University of Utah Health Sciences Center, Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with cystic fibrosis (CF) and exocrine pancreatic insufficiency (EPI) were recruited from centers with CF specialists.
Pre-assignment Details: Out of 36 participants who entered the screening period (11 days), and treated with Ultrase® MT20, 31 were randomized to first intervention period.
Groups:
- Ultrase® MT20 First, Then Placebo: Ultrase® MT 20 capsules containing enteric-coated minitablets orally daily at a dose stabilized during the first stabilization period (4 days), as per investigator's discretion, for 6 to 7 days in the first intervention period followed by placebo matched to Ultrase® MT 20 capsules orally daily for 6 to 7 days in the second intervention period. Break period of 3 to 6 days and fixed dose second stabilization period of 4 days was maintained after first intervention period.
- Placebo First, Then Ultrase®MT20: Placebo matched to Ultrase® MT 20 capsules orally daily for 6 to 7 days in the first intervention period followed by Ultrase® MT 20 capsules containing enteric-coated minitablets orally daily at a dose stabilized during the first stabilization period (4 days), as per investigator's discretion, for 6 to 7 days in the second intervention period. Break period of 3 to 6 days and fixed dose second stabilization period of 4 days was maintained after first intervention period.
Period: First Intervention Period
Arm/Group | Ultrase® MT20 First, Then Placebo | Placebo First, Then Ultrase®MT20
Started | 14 | 17
Completed | 14 | 16
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1
Period: Second Intervention Period
Arm/Group | Ultrase® MT20 First, Then Placebo | Placebo First, Then Ultrase®MT20
Started | 14 | 16
Completed | 12 | 14
Not Completed | 2 | 2
Not completed — Adverse Event | 2 | 0
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal of consent | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all randomized participants.
Groups:
- Entire Study Population: Includes all participants who received Ultrase® MT20 first and placebo first.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.6 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 20

OUTCOME MEASURES:

1. Primary Outcome: Percent Coefficient of Fat Absorption (CFA)
Description: Percent (%) CFA was calculated as ([fat intake - fat excretion]/fat intake)*100, determined by the stools collected during the 72-hour period which could extend to 96 hours during both intervention periods. Mean CFA percent was calculated for 72-hour/96-hour period during Day 3 to Day 7 in the first and second intervention periods.
Time Frame: Day 3 to Day 7 in first intervention period and second intervention period
Population: Intent-to-Treat (ITT) population included all randomized participants. Here, 'N' (number of participants analyzed) signifies those participants who were evaluated for this outcome measure.
Measure: Mean (Standard Deviation); unit: Percent CFA
Arm/Group | Ultrase® MT20 | Placebo
Number analyzed (Participants) | 25 | 27
Percent CFA | 88.55 (4.94) | 55.61 (25.10)
Statistical Analysis 1: Comparison: Ultrase® MT20 vs Placebo; P-values are from a semi-parametric mixed model on ranked CFA% values including sequence, period, and treatment group as fixed effects; participant identification (ID) as random effect; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Net) = 34.74

2. Secondary Outcome: Percent Coefficient of Nitrogen Absorption (CNA)
Description: Percent (%) CNA was calculated as [(nitrogen intake-nitrogen excretion)/nitrogen intake]*100, determined by the stools collected during the 72-hour period which could extend to 96 hours during both intervention periods. Nitrogen intake was calculated as protein intake/6.25. Mean percent CNA was calculated for 72-hour/96-hour period during Day 3 to Day 7 in the first and second intervention periods.
Time Frame: Day 3 to Day 7 in first intervention period and second intervention period
Population: ITT population included all randomized participants. Here, 'N' (number of participants analyzed) signifies those participants who were evaluated for this outcome measure.
Measure: Mean (Standard Deviation); unit: Percent CNA
Arm/Group | Ultrase® MT20 | Placebo
Number analyzed (Participants) | 25 | 27
Percent CNA | 84.05 (7.24) | 58.78 (20.57)
Statistical Analysis 1: Comparison: Ultrase® MT20 vs Placebo; P-values are from a semi-parametric mixed model on ranked CNA% values including sequence, period, and treatment group as fixed effects, and participant ID as random effect; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 25.68

3. Other Pre Specified Outcome: Number of Bowel Movements
Description: Number of bowel movements of each participant was calculated from frequency of stools by the participant per day. Mean daily number of bowel movements on Day 3 for the first treatment period and second treatment period was summarized.
Time Frame: Day 3 on first intervention period and second intervention period
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: bowel movements
Arm/Group | Ultrase® MT20 | Placebo
Number analyzed (Participants) | 29 | 30
bowel movements | 1.5 (1.0) | 3.1 (1.8)

4. Other Pre Specified Outcome: Percentage of Stool Categorized by Consistency
Description: Stool consistency was categorized as hard, formed/normal, soft or watery stool. Percentage of stools of a specific consistency of each participant was calculated as the number of stools with a specific consistency relative to the total number of stools during the collection period. Mean percentage of stool with specific consistency on Day 4 for the first treatment period and second treatment period period for total participants was summarized.
Time Frame: Day 4 on first intervention period and second intervention period
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of stools
Arm/Group | Ultrase® MT20 | Placebo
Number analyzed (Participants) | 28 | 28
percentage of stools
  Hard Stools | 11.31 (27.98) | 3.57 (18.90)
  Formed/Normal Stools | 76.19 (39.13) | 25.71 (43.84)
  Soft Stools | 12.50 (29.27) | 66.73 (45.08)
  Watery Stools | 0 (0) | 3.99 (13.65)

ADVERSE EVENTS:
Time Frame: Day 1 of first stabilization period up to Day 7 of second intervention period
Description: Adverse event (AE) was defined as any untoward medical occurrence regardless of causal relationship to study medication. Serious adverse event (SAE) was any event that resulted in death, life threatening, required or prolonged in-patient hospitalization, significant disability/incapacity,or was a congenital anomaly/birth defect.
Groups:
- Ultrase® MT20: Ultrase® MT 20 capsules containing enteric-coated minitablets orally daily at a dose stabilized during the first stabilization period (4 days), as per investigator's discretion,for 6 to 7 days in either first intervention period or second intervention period.
Arm/Group | Ultrase® MT20 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/30 | 1/31
Other Adverse Events (participants affected / at risk) | 17/30 | 27/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ultrase® MT20 (N=30) | Placebo (N=31)
General physical health deterioration (General disorders) | 0 | 1 — All SAEs reported in this table were unrelated to study drug and all occurred in the same subject.
Pyrexia (General disorders) | 0 | 1
Breath sounds abnormal (Investigations) | 0 | 1
Pulmonary function test decreased (Investigations) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ultrase® MT20 (N=30) | Placebo (N=31)
Abdominal pain (Gastrointestinal disorders) | 2 | 12
Abdominal pain upper (Gastrointestinal disorders) | 4 | 6
Constipation (Gastrointestinal disorders) | 2 | 2
Flatulence (Gastrointestinal disorders) | 1 | 5
Alaninie aminotransferase increased (Investigations) | 1 | 2
Fecal fat increased (Investigations) | 4 | 9
Weight decreased (Investigations) | 0 | 3
Abdominal tenderness (Gastrointestinal disorders) | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 3
Nausea (Gastrointestinal disorders) | 0 | 5
Vomiting (Gastrointestinal disorders) | 0 | 3
Blood glucose increased (Investigations) | 0 | 2
Laboratory test abnormal (Investigations) | 3 | 7
Headache (Nervous system disorders) | 2 | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Rales (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Decreased appetite (Metabolism and nutrition disorders) | 0 | 2
Epistaxis (Vascular disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Restrictions may vary in accordance with each agreement that is negotiated with individual investigators. Sponsor will allow publication after multi-center publication has been published or after an agreed period of time if no such multi-center publication is submitted for publication. Sponsor can ask that Sponsor's confidential information be removed from any publication and defer publication for period of time to allow Sponsor to obtain patent or other intellectual property right protection.